CLINICAL TRIAL: NCT05065749
Title: Clinical Results of Asqelio Trifocal Diffractive Intraocular Lens
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASQT012021
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Cataract
Keywords: cataract surgery; intraocular lens; multifocal refractive correction
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate the clinical outcomes six months after implantation of the trifocal diffractive intraocular lens Asqelio Trifocal IOL TFLIO130C in healthy subjects submitted to non-traumatic cataract surgery.

This clinical performance will be assessed in terms of refractive error, visual performance at different distances, incidence of adverse events and complications following implantation, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to cataract surgery and implanted with Asqelio Trifocal IOL TFLIO130C
* Patients signing a consent form
* Patients seeking spectacle-independence following surgery
* IOL power between +5.00 and +34.00 D
* Transparent intraocular media, except for the cataract prior to surgery, in both eyes
* Postoperatory potential visual acuity of 20/25 or better.

Exclusion Criteria:

* Preoperatory corneal astigmatism greater than 0.75D
* Patients not providing informed consent
* Previous corneal surgery or trauma
* Irregular cornea (i.e. keratoconus)
* Choroidal hemorrhage
* Microophthalmos
* Severe corneal dystrophy
* Uncontrolled or medically controlled glaucoma
* Clinically significant macular changes
* Severe concomitant ocular disease
* Not age-related cataract
* Severe optic nerve atrophy
* Diabetic retinopathy
* Ambyopia
* Extremely shallow anterior chamber
* Severe chronic uveitis
* Pregnant or lactating
* Rubella
* Mature/Dense cataract sifficulting preoperative fundus assessment
* Previous retinal detachment
* Concurrent participation in other investigation using drugs or clinical devices
* Expecting ocular surgery within the study period

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 50 years of age or older submitted to cataract surgery and implanted with the Asqelio Trifocal IOL TFLIO130C according to regular clinical practice
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Six months after implantation
  Percentage of subjects with adverse events (Ocular and Not Ocular, Severe and Not Severe), including secondary surgical procedures
Refraction | Six months after implantation
  Manifest refraction both monocular and binocularly using subjective methods

SECONDARY OUTCOMES:
Uncorrected visual acuity for distance (4m) | Six months after implantation
  Monocular visual acuity for distance (4m), without any additional correction, using ETDRS vision chart
Best-corrected visual acuity for distance (4m) | Six months after implantation
  Monocular visual acuity for distance (4m), with the best correction for distance, using ETDRS vision chart
Uncorrected visual acuity for intermediate | Six months after implantation
  Monocular visual acuity for intermediate distance (60cm), without any additional correction, using ETDRS vision chart
Best-corrected visual acuity for intermediate | Six months after implantation
  Monocular visual acuity for intermediate distance (60cm), with the best correction for distance, using ETDRS vision chart
Uncorrected visual acuity for near | Six months after implantation
  Monocular visual acuity for near distance (40cm), without any additional correction, using ETDRS vision chart
Best-corrected visual acuity for near | Six months after implantation
  Monocular visual acuity for near distance (40cm), with the best correction for distance, using ETDRS vision chart
Contrast sensitivity function (CSF) | Six months after implantation
  CSF with best correction, with and without induced glare, using the Clinical Trial Suite
Defocus curve | Six months after implantation
  Defocus curve of visual performance varying the stimulus vergence from -4.0 D to +1.0 D in 0.5 D steps with the best correction for distance

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - OftalVist Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - OftalVist Alicante, Alicante

REFERENCES:
- [Derived] Tana-Rivero P, Tana-Sanz P, Tana-Sanz S, Montes-Mico R, Cervino A. Recognition vs resolution charts for defocus curve determination in trifocal intraocular lenses. J Cataract Refract Surg. 2024 Sep 1;50(9):942-946. doi: 10.1097/j.jcrs.0000000000001491. PMID 38780434